CLINICAL TRIAL: NCT04956120
Title: Effect of Citrate Dialysate on Vascular Calcification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Fresenius Medical Care Renal Therapies Group (FMCRTG) (Unknown)
Responsible Party: Principal Investigator, Charles O'Neill, Professor, Emory University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00002119
Record Dates: First submitted 2021-06-30; First posted 2021-07-09 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Vascular Calcification
Keywords: Hemodialysis; Breast arterial calcification
MeSH Terms: conditions — Vascular Calcification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Citrate Dialysate then Standard Dialysate (Experimental): Participants receiving hemodialysis using a citrate acid concentrate dialysate for the first year of the study, then receiving hemodialysis using a non-citrate acid concentrate dialysate (standard dialysate) for the second year of the study.
  Interventions: Device: Citrate Dialysate; Device: Standard Dialysate
- Standard Dialysate then Citrate Dialysate (Active Comparator): Participants receiving hemodialysis using a non-citrate acid concentrate dialysate for the first year of the study, then receiving hemodialysis using a citrate acid concentrate dialysate for the second year of the study.
  Interventions: Device: Citrate Dialysate; Device: Standard Dialysate

INTERVENTIONS:
Device: Citrate Dialysate — Dialysate is generated during dialysate from two concentrates (acid concentrate and bicarbonate concentrate) mixed with treated water. When used, citrate is provided in the acid concentrate. The acid concentrate with citrate is approved for this use by the FDA and will be used according to standard procedures without altered dialysis machine settings.
  Other Names: Citrasate
Device: Standard Dialysate — Dialysate is generated during dialysate from two concentrates (acid concentrate and bicarbonate concentrate) mixed with treated water. The acid concentrate without citrate is approved for this use by the FDA and will be used according to standard procedures without altered dialysis machine settings.
  Other Names: Naturalyte

SUMMARY:
The goal of this study is to determine whether hemodialysis with citrate slows the progression of vascular calcification. Participants will be dialyzed with one of two standard dialysis solutions, one with and one without citrate, for 12 months and then switched to the other solution for 12 months. Vascular calcification will be measured on mammograms that will be performed at 6-month intervals and additional blood samples will be obtained at 6-month intervals.

DETAILED DESCRIPTION:
Vascular calcification is a significant problem in dialysis patients that leads to poor outcomes. Currently there is no therapy that directly addresses this problem. Some of the dialysis solutions (dialysates) currently in use contain citrate, a potent inhibitor of calcium precipitation. In particular, citrate can bind to nascent hydroxyapatite crystals and prevent their propagation. Blood citrate levels are greater after dialysis with citrate dialysates than with non-citrate dialysates, which could slow vascular calcification. However, this has never been investigated. Prior research has shown that arterial calcification can be easily detected and reliably measured on routine digital mammograms, with sufficient sensitivity to follow progression. Mammography is more sensitive in detecting arterial calcification than other imaging and associated with far less radiation and cost. This will allow the researchers to detect differences between citrate and non-citrate dialysates in a safe and convenient way. Participants will be dialyzed with one of two standard dialysis solutions, one with and one without citrate, for 12 months and then switched to the other solution for 12 months. Vascular calcification will be measured by mammography every 6 months. The endpoint will be the difference in the rate of progression of breast arterial calcification (BAC) between dialysis with citrate and non-citrate dialysates.

ELIGIBILITY:
Inclusion Criteria:

* hemodialysis patients with BAC on mammograms

Exclusion Criteria:

* current warfarin use
* severe hyperparathyroidism (likely to undergo parathyroidectomy in the next 2 years)
* difficulty controlling serum calcium (likely to require changes in dialysate calcium concentration in the next 2 years)
* life expectancy < 2 years
* prisoners
* inability to give consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2025-03-18 (Actual); Study Completion 2025-03-18 (Actual)

PRIMARY OUTCOMES:
Length of Calcified Artery Segments | Month 0 (baseline), Month 6, Month 12, Month 18, Month 24
  Rate of progression of breast arterial calcification (BAC) is calculated by linear regression of 3 mammograms in each treatment arm (Months 0, 6 and 12 versus Months 12, 18 and 24). Progression of calcification is quantified as the length of calcified artery segments, measured in millimeters.

CONTACTS AND LOCATIONS:
Overall Officials: W. Charles O'Neill, MD, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Emory Dialysis at Northside, Atlanta, Georgia
  - Emory Dialysis at Greenbriar, Atlanta, Georgia
  - Emory Dialysis at North Decatur, Decatur, Georgia
  - Emory Dialysis at Candler, Decatur, Georgia

IPD SHARING:
Plan to Share IPD: No